CLINICAL TRIAL: NCT03485274
Title: Substance Misuse To Psychiatric Disorders for Cannabis (SToP-C)--an Early Assertive Pharmacotherapy Intervention Pilot Study
Brief Title: Substance Misuse To Psychiatric Disorders for Cannabis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SToP-C
Record Dates: First submitted 2018-03-14; First posted 2018-04-02 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Cannabis Use Disorder; Depressive State; Anxiety State; Depression; Anxiety Disorders; Pharmacotherapy
Keywords: Cannabis; depression; anxiety; medication
MeSH Terms: conditions — Depression; Anxiety Disorders; Marijuana Abuse | interventions — Vortioxetine; Therapeutics

STUDY DESIGN:
Intervention Model Description: prospective randomised single-blinded
Who Masked: Outcomes Assessor
Masking Description: treatment in each intervention arms is masked to the outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vortioxetine Arm (Active Comparator): Oral: 5-20mg daily
  Interventions: Drug: Vortioxetine
- Treatment as Usual (Active Comparator): Any medication or Rx other than vortixoetine
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Drug: Vortioxetine — oral medication taken once daily
  Arms: Vortioxetine Arm
Other: Treatment as Usual — Any pharmacological or non-pharmacotherapy modalities other than use of vortioxetine
  Arms: Treatment as Usual

SUMMARY:
With the recent availability of vortioxetine, and the surging phenomenon of cannabis misuses amongst young abusers, it is a timely opportunity to conduct an early pharmacotherapy intervention study to offer an evidence-based strategy aiming to stop individuals with cannabis use disorders with depressive or anxiety symptoms, to develop into a more chronic disabling dependence or co-morbid state.

ELIGIBILITY:
Inclusion Criteria:

• Cannabis use disorder with anxiety or depressive symptoms or disorders; or positive cannabis test results in 1 month with anxiety or depressive symptoms

Exclusion Criteria:

* Age <16 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed to have Intellectual Disabilities (DSM-5) or Mental Retardation
* Had history of primary psychotic episode
* Had been diagnosed to have substance-induced mood disorder, other than cannabis
* Had been diagnosed to have mood disorders or anxiety disorders
* Had been taking maintenance therapeutic dose of antidepressant continuously >= 6 months AND with depressive symptom or anxiety symptom being in remission
* Had known hypersensitivity to vortioxetine
* Had known history of serotonin syndrome
* Pregnant
* Mother currently breast-feeding
* Currently taking warfarin and/or having poorly controlled bleeding disorder
* Had history of prolonged QTc ≥500ms and/or known unstable or untreated cardiology disease

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
change in severity of Cannabis Use Disorder (CUD) | 6 months
  Change in severity of the cannabis use disorder for the 2 arms as defined by DSM-5

SECONDARY OUTCOMES:
prevalence of Cannabis induced mood disorder | 6 months
  The prevalence of the cannabis induced disorder in both arms
Change in Hamilton anxiety (HAM-A) rating scale | 6 months
  To assess the change of anxiety severity of the two treatment arms using HAM-A for both treatment arms with cut-off of defining anxiety >=14
Change in Hamilton depression (HAM-D) rating scale | 6 months
  To assess the change of depression severity of the two treatment arms using HAM-D for both treatment arms with cut-off of defining depression >=8
Change in cognitive outcome | 6 months
  To assess the change in cognitive outcome using Frontal Assessment Battery in the two treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Albert KK Chung, MBBS(HK), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong